CLINICAL TRIAL: NCT01036243
Title: Tolerance of a Slightly Hydrolyzed Starter Formula Containing Probiotics
Brief Title: Digestive Tolerance of Slightly Hydrolyzed Starter Infant Formula With Probiotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07.06 INF
Record Dates: First submitted 2009-12-17; First posted 2009-12-21 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Infant Nutrition
Keywords: digestive tolerance; night sleep; crying; growth
MeSH Terms: conditions — Crying | interventions — Aging

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Test formula 1 (Experimental): Hydrolyzed formula with probiotics
  Interventions: Dietary Supplement: test formula 1
- test formula 2 (Active Comparator): acidified hydrolyzed formula.
  Interventions: Dietary Supplement: test formula 2
- Test formula 3 (Active Comparator): hydrolyzed formula without probiotics
  Interventions: Dietary Supplement: test formula 3
- reference product (Active Comparator): standard infant formula
  Interventions: Dietary Supplement: reference formula

INTERVENTIONS:
Dietary Supplement: test formula 1 — hydrolyzed formula with probiotics
  Other Names: for 0-6 months as per standard requirement
  Arms: Test formula 1
Dietary Supplement: test formula 2 — acidified hydrolyzed formula
  Other Names: suitable for 0-6 months as per standard requirement
  Arms: test formula 2
Dietary Supplement: test formula 3 — hydrolyzed formula without probiotics
  Other Names: suitable for 0-6 months of age as per standard requirement
  Arms: Test formula 3
Dietary Supplement: reference formula — standard infant formula
  Other Names: suitable for 0-6 months of age as per standard requirement
  Arms: reference product

SUMMARY:
To demonstrate that infants have improved gut comfort when fed a slightly hydrolyzed starter formula containing probiotics compared to infants fed a control hydrolyzed and referenced non-hydrolyzed formula.

DETAILED DESCRIPTION:
Infants often experience undesirable gastrointestinal effects, such as constipation, flatulence. These symptoms are often perceived by the parents as being related to the diet (formula) the baby is consuming. In another hand, infantile colic or fussing/crying is one of the most commonly encountered problems within the first three months of life. The etiology of the disorder remains unknown however, three main theories have been proposed to explain its origin: (i) psychological: due to inadequate mother-infant interaction (ii) gastrointestinal: such as hypertonicity and immaturity of the GI tract and Dietary factors that may influence the stool pattern in formula fed infants are (iii) allergic: due to a reaction against cow's milk protein or other food constituents. e.g. the protein source, the iron content, hydrolyzation of the protein, or the fat source.

It has been reported that infants receiving a casein predominant formula had less unformed stools than those receiving a whey predominant formula. Hydrolysation of protein resulted in reduced gastro-intestinal transit time and some studies using extensively hydrolyzed protein formula have shown more liquid stools.

A reduction of crying hours was also described in infant receiving an hydrolyzed formula. Some probiotics were reported with potential benefit on the gut comfort.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants, 0-1 month old at point of enrollment
* Birth weight < 2500g and > 4500g
* Gestational age < 37 weeks and > 42 weeks
* Infants who cannot be breastfed because of the maternal status
* Willing to exclusively consume the assigned study formula with whey protein
* Are likely to be compliant
* Mother/caregiver demonstrates an understanding of the given information and ability to record the requested data

Exclusion Criteria:

* Congenital illness or malformation
* Significant pre-natal and/or post-natal disease
* Receiving systemic antibiotic treatment at time of enrolment
* Infant with symptoms of allergy to cow's milk
* Infant's family cannot be expected to comply with treatment (feeding regimen)
* Subjects who cannot be expected to comply with treatment
* Currently participating or having participated in another clinical trial during the last month

Ages: 11 Days to 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 480 (Actual)
Dates: Start 2009-12; Primary Completion 2012-01 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
incidence of crying/fussing from 1 to 3 months. | 3 months

SECONDARY OUTCOMES:
growth and night sleep | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: A/Prof. Boosba Vivatvakin, MD, Principal Investigator — Pediatric Gastroenterology Unit,Faculty of Medicine, Chulalongkorn University
Locations (1):
- Chulalongkorn University, Bangkok, Thailand